CLINICAL TRIAL: NCT05465252
Title: Effect of Krill Oil Supplementation on Dry Age-Related Macular Degeneration: A Randomized Controlled Trial
Brief Title: Effect of Omega-3 Fatty Acid Supplementation on Dry-AMD Progression
Acronym: OMEGA-AMD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaodong Sun, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SXD20220608
Record Dates: First submitted 2022-06-09; First posted 2022-07-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Age-Related Macular Degeneration
Keywords: dry age-related macular degeneration; krill oil
MeSH Terms: conditions — Macular Degeneration | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- krill oil (Experimental)
  Interventions: Dietary Supplement: Krill Oil
- olive oil (Placebo Comparator)
  Interventions: Dietary Supplement: Olive Oil

INTERVENTIONS:
Dietary Supplement: Krill Oil — Qualified subjects start to take supplementation from Day 1 in the trial. Specifically, subjects from Intervention group take 4 capsules of krill oil per day.
  Other Names: Superba Boost
  Arms: krill oil
Dietary Supplement: Olive Oil — Qualified subjects start to take placebo from Day 1 in the trial. Specifically, subjects from placebo group take 4 capsules of olive oil, which has the same color and smell as the krill oil.
  Arms: olive oil

SUMMARY:
This randomized, double-blind, placebo-controlled study aims to evaluate the effect of krill oil supplementation in patients with dry age-related macular degeneration (AMD). Participants will receive 4 capsules of krill oil or placebo daily for a period of 3 months. Outcomes will be evaluated after 3-month treatment to assess differences between the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with dry AMD at an early or intermediate stage, classified according to the Beckman Classification and confirmed by fundus photography: (1) Early AMD: medium drusen (>63 μm and ≤125 μm) without AMD-related pigmentary abnormalities; (2) Intermediate AMD: large drusen (>125 μm), with or without AMD-related pigmentary abnormalities.
* Willing to stop supplementation of omega-3 fatty acids, choline, or astaxanthin.
* Willing to sign the informed consent, and willing to attend follow-up visits for at least 3 months.

Exclusion Criteria:

* Any eye with disease that would interfere with the fundus examinations.
* Eye with choroidal neovascularization (CNV), geographic atrophy (GA), or high myopia.
* Surgeries that may interfere with AMD evaluation.
* Long-term use of any medications that are associated with retinal or neural toxicities.
* History of supplementation with lutein, zeaxanthin, DHA, or EPA, unless a wash-out period of at least 8 weeks is completed prior to enrollment.
* Intraocular pressure more than 26 mmHg.
* Received cataract surgery in 3 months.
* Other conditions: subjects with severe systemic diseases; any condition that causes high risk of drop-out, or low compliance, for instance cognition disorder; have been involved in other trial that interfere with the current visit plan; taking other angiogenesis Inhibitors drugs for treating cancer.
* Other conditions not suitable for the current study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Macular Drusen Volume | From enrollment to the end of follow-up at 3 months.
  Macular drusen volume will be quantified using spectral-domain optical coherence tomography (SD-OCT). Automated segmentation of Bruch's membrane and the retinal pigment epithelium (RPE), followed by manual verification, will be performed to calculate drusen volume at baseline and after 3 months of intervention at the same retinal location.
  Change in macular drusen volume will be defined as the percentage change from baseline, calculated as the difference between post-intervention and baseline drusen volume divided by the baseline drusen volume.

SECONDARY OUTCOMES:
Change in Maximum Macular Drusen Height | From enrollment to the end of follow-up at 3 months.
  Maximum macular drusen height will be measured using SD-OCT at baseline and after 3 months of intervention.
  Change in maximum macular drusen height will be defined as the percentage change from baseline, calculated as the difference between post-intervention and baseline maximum drusen height divided by the baseline maximum drusen height.
Change in Best-Corrected Visual Acuity | From enrollment to the end of follow-up at 3 months.
  Best-corrected visual acuity (BCVA) will be assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart and quantified as the total number of letters correctly identified by the participant.
  Change in BCVA will be defined as the absolute change in ETDRS letters from baseline, calculated as the difference between post-intervention and baseline measurements.
Change in Self-Reported Visual Function | From enrollment to the end of follow-up at 3 months.
  Self-reported visual function will be assessed using the 25-item National Eye Institute Visual Function Questionnaire (NEI VFQ-25).
  Change in self-reported visual function will be defined as the absolute change in NEI VFQ-25 total score from baseline, calculated as the difference between post-intervention and baseline scores.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Sun, PHD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No